CLINICAL TRIAL: NCT04319250
Title: The Effectiveness Of Ischemic Compression And Instrument Assisted Soft Tissue Mobilization In Trigger Point Treatment In Patients With Rotator Cuff Tear
Brief Title: The Effectiveness Of Ischemic Compression And IASTM In Trigger Point Treatment In Patients With Rotator Cuff Tear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, Büşra Aksan Sadıkoğlu, Principal Investigator (MSc), Istanbul Aydın University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Büşra Aksan Sadıkoğlu
Record Dates: First submitted 2020-03-19; First posted 2020-03-24 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Rotator Cuff Tears; Shoulder Pain; Myofascial Trigger Point Pain
Keywords: ischemic compression; instrument assisted soft tissue mobilization; trigger point
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Pain; Myofascial Pain Syndromes | interventions — Acupressure; Rehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Ischemic compression and rehabilitation program applied to the group 1
  Interventions: Other: ischemic compression; Other: Rehabilitation Program
- Group 2 (Active Comparator): IASTM and rehabilitation program applied to the group 2
  Interventions: Other: IASTM; Other: Rehabilitation Program

INTERVENTIONS:
Other: ischemic compression — ATNs detected in a total of 13 muscles around the shoulder were applied constant pressure at the level of pain tolerated with the thumb (discomfort severity level 7 to 8 out of 10) and for 90 seconds. This method was applied twice a week for 6 weeks.
  Arms: Group 1
Other: IASTM — In order to apply EDYDM in the treatment of ATN, titanium plated stainless steel was divided into two parts, front and back, with two tools. The sweep was applied to the anterior muscle fibers at an angle of 45 ° for 40 seconds.
  For each TN, continuous pressure was applied with swivel movement at tolerable pain level (discomfort severity level 7 to 8 out of 10) for 1 minute. The back group muscles were applied in the same way.
  Arms: Group 2
Other: Rehabilitation Program — A rehabilitation program consisting of exercises and manual therapy used in the conservative treatment of rotator cuff tear for both groups was applied twice a week for 6 weeks.

SUMMARY:
The aim of this study is to determine the effects of ischemic compression and IASTM techniques on pain, EHA, functionality, anxiety and depression in patients with the diagnosis of RM tear and presence of ATN. In addition, ischemic compression and EDYDM methods were aimed to compare and to reveal which application would be more useful.

DETAILED DESCRIPTION:
In this study participants were randomly divided into two groups. While ischemic compression was applied to one group for the determined active trigger points, instrument assisted soft tissue mobilization (IASTM) was applied to the other group for active trigger points. In addition to the treatment, both groups were subjected to a joint rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Being between 40-65 years old
* Having been diagnosed with partial RM rupture
* RM rupture in MRI image
* At least 3 ATNs in the shoulder complex
* Hawkins-Kennedy and Empty Can tests positive Symptoms for at least 3 months

Exclusion Criteria:

* Sensory problems in the back and shoulders,
* Shoulder instability
* Osteoarthritis in the shoulder joint area
* Glenoid or bone fracture
* Frozen shoulder pathology
* Massive RM rupture
* Rheumatological joint problems
* Shoulder surgery history

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH) | Change from Baseline at 6 weeks
  This is a questionnaire that identifies both functionality and symptoms that can be used in arm, elbow and hand problems. High scores of individuals mean that functional dysfunction is high. Ratings are made between 0 and 100.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | Change from Baseline at 6 weeks
  The levels of pain felt at rest / activity / night were measured using Visual Analogue Scale (VAS).
Shoulder Range of Motion (ROM) | Change from Baseline at 6 weeks
  EHA evaluations of flexion, abduction, internal rotation and external rotation of the shoulder joint were performed in the supine position using the universal goniometer.
Active trigger points | Change from Baseline at 6 weeks
  Active trigger points were evaluated by palpation method according to Travell and Simons criteria. Scalene, upper trapezius, levator scapula, supraspinatus, infraspinatus, subskapularis, teres minor, teres major, deltoid anterior and posterior group fibers, pectoralis major, pectoralis minor, biceps brachii muscles were evaluated with palpation method in terms of trigger point presence.
Pain Pressure Threshold (PPT) | Change from Baseline at 6 weeks
  Wagner Force One ™ FDIX" digital algometer was used to evaluate the pain threshold. Measurements were recorded in kg / cm².
The American Shoulder and Elbow Surgeons Standardized Shoulder Assesment Form (ASES) | Change from Baseline at 6 weeks
  This score consists of 1 questioning pain and 10 questions questioning daily life activities.The total score is at least 0 and at most 100, and the high scores are positively correlated with the normal function.
Emotional state | Change from Baseline at 6 weeks
  The emotional states of the cases were evaluated using the Hospital Anxiety and Depression Scale (HAD), which consists of 14 questions. (HAD). This scale has a 7-question anxiety (HAD-A) subscale that evaluates the anxiety state, and a 7-question depression (HAD-D) subscale that evaluates the state of depression, and a four-point likert scale is used to answer the questions. For the total score of each sub-score, 0-7 points are normal, 8-10 points are at the border, and 11 points are defined as abnormal
Global Rating of Change (GRC) scale | After 6 weeks treatment
  Patient Satisfaction was assessed Global Rating of Change (GRC) scale. The scale used included 5 points (-2: I am much worse. -1: I am worse, 0: I am the same, +1: I am better, +2: I am much better).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydin University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided